CLINICAL TRIAL: NCT05502367
Title: An Open-Label Single and Multiple-dose, Study to Evaluate Safety, Tolerability and Efficacy of ABI-2280 Vaginal Insert (Previously Referred to as ABI-2280 Vaginal Tablet) in Participants With Cervical Squamous Intraepithelial Lesions
Brief Title: A Study of ABI-2280 Vaginal Insert (Previously Referred to as ABI-2280 Vaginal Tablet) in Participants With Cervical Intraepithelial Neoplasia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Antiva Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABI-2280-303
Record Dates: First submitted 2022-08-07; First posted 2022-08-16 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Mutagenesis, Insertional

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Cohort A1: Single and multiple doses of ABI-2280 (Experimental)
  Interventions: Drug: ABI-2280 Vaginal Tablet/Insert
- Cohort A2: Multiple doses of ABI-2280 (Experimental)
  Interventions: Drug: ABI-2280 Vaginal Tablet/Insert
- Cohort A3: Multiple doses of ABI-2280 (Experimental)
  Interventions: Drug: ABI-2280 Vaginal Tablet/Insert
- Cohort A4: Multiple doses of ABI-2280 (Experimental)
  Interventions: Drug: ABI-2280 Vaginal Tablet/Insert
- Cohort A5: Multiple doses of ABI-2280 (Experimental)
  Interventions: Drug: ABI-2280 Vaginal Tablet/Insert
- Cohort A6: Multiple doses of ABI-2280 (Experimental)
  Interventions: Drug: ABI-2280 Vaginal Tablet/Insert
- Cohort A7: Multiple doses of ABI-2280 (Experimental)
  Interventions: Drug: ABI-2280 Vaginal Tablet/Insert
- Cohort A8: Intermittent multiple doses of ABI-2280 (Experimental)
  Interventions: Drug: ABI-2280 Vaginal Tablet/Insert
- Cohort A9: Multiple doses of ABI-2280 (Experimental)
  Interventions: Drug: ABI-2280 Vaginal Tablet/Insert

INTERVENTIONS:
Drug: ABI-2280 Vaginal Tablet/Insert — Vaginal Tablet

SUMMARY:
This is an open-label study to evaluate the safety, tolerability, and efficacy of ABI-2280 in participants with cervical squamous intraepithelial lesions. This study is divided into 2 parts - Part A and Part B.

Part A consists of up to 9 dose escalation cohorts. Part B consists of dose expansion cohorts.

Participants will self-administer ABI-2280.

ELIGIBILITY:
Inclusion Criteria:

* Women, 25 to 55 years old.
* For Cohorts A1 and A2 in Part A, participants with biopsy-confirmed CIN (with visible lesions) regardless of p16 positivity may be enrolled upon consultation with PI and Medical Monitor. These participants will not be required to get LLETZ if not medically necessary, as determined by the PI in consultation with the Medical Monitor.
* For Cohorts A3 and above in Part A and Part B POC cohorts, biopsy-confirmed cHSIL that is p16+ (p16INK4a expressed) within 60 days of enrollment (dosing) with no evidence of invasive cancer in any specimen. If biopsy was performed ≥ 60 days before planned enrollment, participants must agree to have another biopsy performed at the Screening visit, unless approved by the Medical Monitor.
* A positive high-risk HPV (hrHPV) result by provider-obtained cervical swab at screening or previously obtained and documented within the past 3 months.
* No prior treatment for Cervical intraepithelial neoplasia (CIN).
* Generally, in good health with no clinically significant pulmonary, cardiac, gastro-enterologic, neurologic, renal, musculoskeletal, rheumatologic, metabolic, neoplastic, or endocrine disease.

Exclusion Criteria:

* Women who are pregnant, plan to become pregnant in the next 4 months, or lactating females.
* Unwilling to use stringent methods of contraception (including barrier method, as well as another acceptable method) throughout the course of the study.
* History of cancer, except basal cell or squamous cell carcinoma of the skin.
* History of genital herpes with outbreak within prior 12 months.
* Have an active pelvic or non-HPV (Human papillomavirus) vaginal infection (e.g., that was detected by a positive urine screen for gonorrhea or chlamydial infection, bimanual exam consistent with pelvic inflammatory disease, positive bedside testing criteria for bacterial vaginosis, candida vaginitis or trichomonal vaginitis, etc).
* Current or recent abnormal vaginal discharge and /or abnormal vaginal bleeding.
* Had a therapeutic abortion or miscarriage less than 3 months prior.
* Any clinically significant immune suppressing condition.
* Participants with a significant acute condition or any other condition that in the opinion of the Investigator might interfere with the evaluation of the study objectives.
* Women who, in the PI's judgment, would be harmed by the delay in undergoing definitive treatment as a result of study participation and the ABI-2280 Vaginal Tablet dosing schedule.
* Vaccination (even 1 dose) with a prophylactic HPV vaccine (i.e., Gardasil®, Gardasil®-9 or Cervarix®) in the last 3 months.
* Vaccination with a therapeutic HPV vaccine.

  * Other inclusion/exclusion criteria may apply

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-09-10 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (Safety and Tolerability) | From Baseline to Day 42 post dose administration
  For Parts A and B, to assess the safety and tolerability of ABI-2280 Vaginal Tablet by the incidence and severity of Adverse events (AEs).

SECONDARY OUTCOMES:
Histopathologic changes in cHSIL by large loop excision of the transformation zone (LLETZ) speciment | 12 weeks after the first dose of ABI-2280 Vaginal Tablet
  To assess histopathologic changes in cHSIL by LLETZ
Pharmacokinetics of ABI-2280 after single and multiple doses | PK time points will begin on Day 1 and will continue up to Day 49 (depending on the Cohort)
  Pharmacokinetics sampling of ABI-2280 will be taken at various time points after single and multiple doses to assess systemic exposure.

OTHER OUTCOMES:
Exploratory Endpoint | hrHPV testing to occur at baseline up to end of study (Day 84)
  To evaluate the viral clearance of high-risk human papillomavirus (hrHPV)

CONTACTS AND LOCATIONS:
Locations (7):
- East Sydney Doctors, Darlinghurst, New South Wales, Australia
- Peru (2):
  - CerviCusco, Cusco
  - Ginobs S.A., Lima
- South Africa (4):
  - Farmovs, Bloemfontein, Free State
  - Nafasi Integrated Solutions, Sunnyside, Gauteng
  - Botho ke Bontle Health Services, Waltloo, Gauteng
  - Gole Biomedical Research Centre, Ga-Mothapo, Limpopo

IPD SHARING:
Plan to Share IPD: No